CLINICAL TRIAL: NCT00468689
Title: A Two-Part Dose-Rising Study to Evaluate the Safety, Tolerability and Pharmacokinetics of SB-751689 When Administered as an Oral Formulation at Supratherapeutic Dose Levels in Healthy Adult Subjects.
Brief Title: Evaluation Of SB-751689 Administered At Supratherapeutic Dose Levels In Healthy Adult Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CR9107262
Record Dates: First submitted 2007-05-01; First posted 2007-05-03 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-10

CONDITIONS: Osteoporosis
Keywords: SB-751689,; Calcium-sensing receptor antagonist (CaR),; Osteoporosis,; Parathyroid hormone (PTH),; Oral dose
MeSH Terms: conditions — Osteoporosis | interventions — Ketoconazole

INTERVENTIONS:
Drug: SB-751689 oral tablets (100 and 400 ng)
Drug: Ketoconazole (NIZORAL) oral tablets (200 mg)
  Other Names: SB-751689 oral tablets (100 and 400 ng)

SUMMARY:
This study will evaluate the safety, tolerability and exposure of SB-751689 when administered alone at supratherapeutic doses and when SB-751689 is co administered with ketoconazole, a PGP/CYP3A4 inhibitor that increases exposure of SB-751689. Data from this study will enable the planning and conduct of a QTc study for SB-751689.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-60yrs, with BMI of 19-31kg/m2.
* Females must be of non-childbearing potential.
* Subjects must be able to give consent and comply with restrictions of study.

Exclusion Criteria:

* Clinically relevant abnormality from history, physical, 12-lead ECG, Holter monitoring, or clinical laboratory examination.
* Positive urine drug screen.
* Positive urine test for alcohol.
* Contine levels indicative of smoking.
* Positive HIV or Hep B and/or C assay.
* History or smoking in last year or >10 pack/year history of smoking overall.
* History of regular alcohol consumption (7 units/week for women and 14 units/week for men) within 6 months of study.
* History of drug abuse within 6 months of study.
* Participation in another drug trial within 30 days of first dose.
* Exposure to more than 4 new chemical entities within 12 months of first dose.
* Use of prescription and non-prescription drugs including dietary supplements, herbals and St. John's wort within 14 days of first dose.
* Consumption of red wine, grapefruit, grapefruit juice and grapefruit products within 14 days of first dose.
* Donation of blood in excess of 500 mL within 56 days of dosing.
* Evidence of renal, hepatic or biliary impairment.
* History of serious gastrointestinal disease or history of gastrointestinal surgical procedure that might affect absorption of study drug.
* History of sensitivity to any of the study medications.
* History of clinically significant cardiovascular disease.
* History of pernicious anemia, pancreatitis, osteosarcoma or kidney stones. Medical conditions which might alter bone metabolism.
* Liver function tests above ULN at screening and PTH, glucose, and CPK outside the reference range at screening.
* Males unwilling to refrain from fathering a child during the study and for 14 days following the last dose of study medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2007-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of SB-751689 doses determined from clinical safety and tolerability data from all adverse event reporting, 12-lead ECGs, vital signs, nursing/physician observation, and safety laboratory tests | throughout the study

SECONDARY OUTCOMES:
PK and of SB-751689 as determined by AUC, Cmax, tmax, and half-life. PD effects (PTH, serum Ca) as determined by AUC, Emax, tmax, maximum change and % change from baseline, duration of effect, duration above ULN for PTH. | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States